CLINICAL TRIAL: NCT01188733
Title: Hepatic Hemodynamic Responses to Long-acting Octreotide in Patients With Cirrhosis Hepatic Hemodynamic Responses to Long-acting Octreotide in Patients With Cirrhosis
Brief Title: Efficacy of Long-acting Octreotide (Sandostatin LAR) in Reducing Portal Pressure in Patients With Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Patrick S. Kamath, Division of Gastroenterology and Hepatology, Mayo Clinic, Rochester MN 55905
Allocation: Randomized | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-005739
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Cirrhosis; Portal Hypertension; Esophageal Varices
Keywords: portal hypertension; varices; cirrhosis; octreotide; somatostatin analog; Child Pugh Class A,B
MeSH Terms: conditions — Fibrosis; Hypertension, Portal; Esophageal and Gastric Varices; Varicose Veins | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sandostatin LAR 10mg (Experimental): Sandostatin LAR ( long-acting octreotide) administered every 28 days in a dose of 10mg
  Interventions: Drug: Long acting octreotide 10mg
- Sandostatin LAR 30mg (Experimental): Comparison of drug doses
  Interventions: Drug: Long acting Octreotide 30mg
- Saline (Placebo Comparator): Saline control
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Long acting octreotide 10mg — Comparison of different doses
  Other Names: Long-acting octreotide
  Arms: Sandostatin LAR 10mg
Drug: Long acting Octreotide 30mg — Comparison of drug doses
  Arms: Sandostatin LAR 30mg
Drug: Saline — Comparison of drug doses
  Arms: Saline

SUMMARY:
Octreotide is used to control variceal bleeding. However, octreotide has to be given through the vein and is effective for less than two hours.

In this study the investigators determined whether a long-acting preparation of octreotide (Sandostatin LAR)given as an intra-muscular injection every month could decrease portal pressure, and thus be used to prevent variceal bleeding in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis documented by biopsy, or suggested by characteristic features on abdominal imaging (nodular appearance, irregular contour) along with impaired synthetic liver function and thrombocytopenia and Child Turcotte Pugh Class A or B.
2. presence of small esophageal varices, defined as varices < 5 mm in diameter, without red signs documented on endoscopy within 3 months of enrollment
3. age ≥ 18 years

Exclusion Criteria:

* pregnant, lactating or of child-bearing potential and not practicing acceptable method of birth control
* allergic to sandostatin
* high risk varices on endoscopy carried out within 3 months of assessment (large varices or red signs)
* Child Turcotte Pugh Class C cirrhosis
* hepatocellular carcinoma
* evidence of ongoing alcohol or illicit drug abuse within 6 months of the study
* serum creatinine greater than 2 mg/dL
* platelet count below 50,000 per microliter
* prothrombin time 4 seconds or more greater than control
* human immunodeficiency virus (HIV) positive
* symptomatic gallstones
* previous history of upper gastrointestinal bleeding in the past 3 months, defined as hematemesis and/or melena
* previous history of variceal bleeding
* history of congestive heart failure , unstable angina, sustained ventricular tachycardia, or ventricular fibrillation
* use of any investigational drug within 1 month prior to screening and
* current use of beta blockers or long-acting nitrates, any other drug therapy known to have an influence on portal pressure (diuretics were allowed provided patients were on a stable dose for at least 30 days).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1998-06; Primary Completion 2000-07 (Actual); Study Completion 2000-12 (Actual)